CLINICAL TRIAL: NCT03030898
Title: Analysis of Respiratory Variations of the Internal Jugular Vein as a Predictor of Fluid Responsiveness During Mechanical Ventilation
Brief Title: Analysis of Respiratory Variations of the Right Internal Jugular Vein as a Predictor of Fluid Responsiveness During Mechanical Ventilation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Military Hospital of Tunis (Other)
Responsible Party: Principal Investigator, Lebbi Anis, Clinical Professor, Military Hospital of Tunis
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 9829260098237333
Record Dates: First submitted 2017-01-19; First posted 2017-01-25 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2017-01

CONDITIONS: Jugular Veins; Ultrasonography

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- respiratory variation of the right internal jugular vein (Other)
  Interventions: Diagnostic Test: respiratory variation of the right internal jugular vein

INTERVENTIONS:
Diagnostic Test: respiratory variation of the right internal jugular vein — respiratory variation of the right internal jugular vein vs respiratory variation of superior and inferior cava vena

SUMMARY:
The idea of this work came during a carotid surgery, when we noticed a respiratory variation of the right internal jugular vein. Also, because of the interest of evaluating the preload dependence during an intervention or reanimation where it is difficult to access the other monitoring methods . The aim of the study was to test the hypothesis that respiratory changes in right internal jugular vein diameter are similar to respiratory changes in superior and inferior vena cava in mechanically ventilated patients and therefore help to predict fluid responsiveness.

ELIGIBILITY:
Inclusion Criteria:

* older than 18 years
* Mechanical Ventilation

Exclusion Criteria:

* no exclusion Criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-04-25 (Estimated); Study Completion 2017-12-28 (Estimated)

PRIMARY OUTCOMES:
Respiratory Variation of the Right Internal Jugular Vein ∆DRIJV | through study completion, an average of 1 year
  Difference (Δ) between the maximum and the minimum diameter value/maximum diameter .
Respiratory Variation of the superior vena cava ∆DSVC | through study completion, an average of 1 year
  Difference (Δ) between the maximum and the minimum diameter value/maximum diameter .

SECONDARY OUTCOMES:
Respiratory Variation of the inferior vena cava ∆DIVC | through study completion, an average of 1 year
  Difference (Δ) between the maximum and the minimum diameter value/minimum diameter .

CONTACTS AND LOCATIONS:
Overall Officials: Anis Lebbi, Study Director — Military Hospital of Tunis; Mejdi Ferjaoui, Principal Investigator — Military Hospital of Tunis; Trabelsi Walid, Study Chair — Military Hospital of Tunis; Abdelkader Ben Gabsia, Study Chair — Military Hospital of Tunis; Emel Rafrafi, Study Chair — Military Hospital of Tunis; Amine Skouri, Study Chair — Military Hospital of Tunis; Kaouther Fares, Study Chair — Military Hospital of Tunis; Walid Sallami, Study Chair — Military Hospital of Tunis; Iheb Labbene, Study Chair — Military Hospital of Tunis; Mustapha Ferjani, Study Chair — Military Hospital of Tunis